CLINICAL TRIAL: NCT03434769
Title: Phase I Clinical Trial of AntiCD19 Chimeric Antigen Receptor T Cells for Treatment of Relapsed or Refractory Non Hodgkin Lymphoma
Brief Title: AntiCD19 Chimeric Antigen Receptor T Cells for Relapsed or Refractory Non Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Benjamin Tomlinson (Other)
Responsible Party: Sponsor-Investigator, Benjamin Tomlinson, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2417
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Cyclophosphamide; Fludarabine; Chimeric antigen receptor T cells
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cyclophosphamide + Fludarabine + Infusion of CAR-T Cells (Experimental): Lymphodepletive regimen, consisting of Cyclophosphamide 60mg/kg IV on day -6 and Fludarabine 25mg/m2 IV on days -5 to -3. Followed by infusion of Chimeric antigen receptor T-cells (CAR-T) on day 0
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: CAR-T Cells

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide 60mg/Kg on day -6
  Other Names: Cytoxan; Endoxan; Neosar; Procytox; Revimmune; Cycloblastin
Drug: Fludarabine — Fludarabine 25mg/m^2 IV on days -5 to -3
  Other Names: Fludara
Biological: CAR-T Cells — Chimeric antigen receptor T cells to be implemented in a "3 + 3" design on day 0
  Level -1 (1 x 105 cells/kg)
  Level 1 [Starting dose] (5 x 105 cells/kg)
  Level 2 (1 x 106 cells/kg)
  Level 3 (2 x 106 cells/kg)

SUMMARY:
The purpose of this study is to determine if it is possible to treat your cancer with a new type of T cell-based immunotherapy (therapy that uses your immune system to treat the cancer). T cells are a type of white blood cell that helps the body fight infections. This treatment uses T cells already present within your body that have been modified outside of the body and returned to target your cancer. This type of treatment is sometimes referred to as adoptive cell transfer (ACT). In this study the specific type of cells that will be used is called chimeric antigen receptor T cells (CAR T cells). Another purpose of this study is to learn about the side effects and toxicities related to this treatment.

DETAILED DESCRIPTION:
Primary Objective: To determine the safety of the treatment of relapsed or refractory B cell lymphomas with chimeric antigen receptor T cells targeting cluster of differentiation antigen 19 (CD19) and to find the recommended phase II dose for this cellular therapy

Secondary Objectives

* To describe the safety profile of the infusion of CAR-T cells targeting CD19.
* To describe the toxicities related to infusion of CAR-T cells targeting CD19.
* To describe the overall response rate and complete response rate of relapsed B cell malignancies treated with CAR-T cells targeting CD19.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have relapsed or refractory non-Hodgkin lymphoma treated with at least two lines of therapy. Disease must have either progressed after the last regimen or presented failure to achieve partial or complete remission with the last regimen.
* The patient's lymphoma must be CD19 positive, either by immunohistochemistry or flow cytometry analysis on the last biopsy available.
* Eastern Cooperative Oncology Group (ECOG) Performance status ≤ 2
* Total bilirubin ≤ 1.5 times the institutional upper limit of normal
* Aspartate transaminase (AST or SGOT) ≤ 3 X institutional upper limit of normal
* Alanine transaminase (ALT or SGPT) ≤ 3 X institutional upper limit of normal
* Serum Creatinine ≤ 2 X the institutional upper limit of normal
* Subjects must have the following hematologic function parameters:

  * absolute neutrophil count (ANC)>1,000/uL
  * Absolute Lymphocyte Count >100/uL
  * Platelets >50,000/uL
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Autologous transplant within 6 weeks of planned CAR-T cell infusion
* History of allogeneic stem cell transplant.
* Recipient of CAR-T cell therapy outside of this protocol.
* Active central nervous system or meningeal involvement by lymphoma. Subjects with untreated brain metastases or central nervous system (CNS) disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with a history of CNS or meningeal involvement must be in a documented remission by cerebrospinal fluid evaluation and contrast-enhanced MRI imaging for at least 90 days prior to registration.
* Active malignancy, other than non-melanoma skin cancer, carcinoma in situ (e.g. cervix, bladder, breast).
* HIV seropositivity
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with the potential for teratogenic or abortifacient effects. Women of child bearing potential must have a negative serum pregnancy test. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAR-T cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study.
* Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on any bone marrow biopsy prior to initiation of therapy
* Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive patients will be excluded.)
* Patients with history of clinically relevant CNS pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease.
* History of autoimmune disease (i.e. rheumatoid arthritis, systemic lupus erythematosus) with requirement of immunosuppressive medication within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2036-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Lymphoma response | Up to 12 months after getting CAR-T infusion
  The 2014 Lugano Response for Malignant Lymphoma will be used the following categories of response: : Complete Response (CR), Partial Response (PR), Stable Disease (SD), Relapse and Progression (PD).

SECONDARY OUTCOMES:
Duration of response | Up to 12 months after getting CAR-T infusion
  This is measured, only in responders, from the documented beginning of response (CR or PR) to the time of relapse.
Disease-free survival | Up to 12 months after getting CAR-T infusion
  Survival is defined as the date of study entry to the date of death. Disease-free survival is measured from the time of occurrence of disease-free state to disease recurrence or death from lymphoma or acute toxicity of treatment.
Disease-specific survival | Up to 12 months after getting CAR-T infusion
  To minimize the risk of bias, the event should be recorded as death from lymphoma, or from toxicity from the drug. Death from unknown causes should be attributed to the drug.
Progression-free survival | Up to 12 months after getting CAR-T infusion
  Progression-free Survival (PFS) is defined as the time from entry onto study until lymphoma progression or death from any cause.
Time to progression | Up to 12 months after getting CAR-T infusion
  Time to progression (TTP) is defined as the time from study entry until lymphoma progression or death due to lymphoma.
Time to treatment failure | Up to 12 months after getting CAR-T infusion
  Time to treatment failure (event-free survival) is measured from the time from study entry to any treatment failure including discontinuation of treatment for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Tomlinson, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- [Derived] Ghobadi A, Caimi PF, Reese JS, Goparaju K, di Trani M, Ritchey J, Jackson Z, Tomlinson B, Schiavone JM, Kleinsorge-Block S, Zamborsky K, Eissenberg L, Schneider D, Boughan KM, Zabor EC, Metheny L, Gallogly M, Kruger W, Kadan M, Worden A S A, Sharma A, Cooper BW, Otegbeye F, Sekaly RP, Wald DN, Carlo-Stella C, DiPersio J, Orentas R, Dropulic B, de Lima M. Treatment of non-Hodgkin lymphoma with point-of-care manufactured CAR T cells: a dual institution, phase 1 trial. EClinicalMedicine. 2025 Mar 4;81:103138. doi: 10.1016/j.eclinm.2025.103138. eCollection 2025 Mar. PMID 40115173
- [Derived] Maschan M, Caimi PF, Reese-Koc J, Sanchez GP, Sharma AA, Molostova O, Shelikhova L, Pershin D, Stepanov A, Muzalevskii Y, Suzart VG, Otegbeye F, Wald D, Xiong Y, Wu D, Knight A, Oparaocha I, Ferencz B, Roy A, Worden A, Kruger W, Kadan M, Schneider D, Orentas R, Sekaly RP, de Lima M, Dropulic B. Multiple site place-of-care manufactured anti-CD19 CAR-T cells induce high remission rates in B-cell malignancy patients. Nat Commun. 2021 Dec 10;12(1):7200. doi: 10.1038/s41467-021-27312-6. PMID 34893603